CLINICAL TRIAL: NCT03860480
Title: Erector Spinae Plane Block For Analgesia Following Video-Assisted Thoracoscopic Surgery : A Multi-Center Randomized Controlled Trial
Brief Title: Erector Spinae Plane Block For Analgesia Following Video-Assisted Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Ariane Clairoux, Assistant Professor Anesthesiology and Pain Medicine, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MP-12-2019-1640
Record Dates: First submitted 2019-01-21; First posted 2019-03-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Thoracic Surgery, Video-Assisted
Keywords: Post-operative analgesia; VATS; Thoracoscopic surgery; Erector spinae plane block; Regional anesthesia
MeSH Terms: interventions — Parapsychology; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Control group : Postoperative patient-controlled analgesia (PCA) pumps with Hydromorphone + Sham Erector Spinae Plane Block Intervention group : Postoperative patient-controlled analgesia (PCA) pumps with Hydromorphone + Erector Spinae Plane Block
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ESP with Bupivacaine 0.5% (Active Comparator): The Erector Spinae Block (ESP) will be performed using the method described by Forero et al and Hamilton et al. in 2017 by an expert regional anesthesiologist.
  Thirty milliliters of bupivacaine at a concentration of 0.5% with epinephrine 1:200 000 will be injected depending on the patient's allocation.
  Patient controlled analgesia (PCA) settings for both groups will remain the same: hydromorphone with a bolus of 0,2 mg, lockout time of 5 minutes and no background infusion. The PCA will be started when the patient is transferred to the postanesthesia care unit (PACU).
  Interventions: Procedure: ESP with Bupivacaine 0.5%
- ESP with Saline 0.9% (Sham Comparator): The Erector Spinae Block (ESP) will be performed using the method described by Forero et al and Hamilton et al. in 2017 by an expert regional anesthesiologist.
  Thirty milliliters of a placebo solution (normal saline) will be injected depending on the patient's allocation.
  Patient controlled analgesia (PCA) settings for both groups will remain the same: hydromorphone with a bolus of 0,2 mg, lockout time of 5 minutes and no background infusion. The PCA will be started when the patient is transferred to the postanesthesia care unit (PACU).
  Interventions: Procedure: ESP with Saline 0.9%

INTERVENTIONS:
Procedure: ESP with Bupivacaine 0.5% — Regional anesthesia procedure with Bupivacaïne 0.5%
  Arms: ESP with Bupivacaine 0.5%
Procedure: ESP with Saline 0.9% — Regional anesthesia procedure with Normal Saline
  Arms: ESP with Saline 0.9%

SUMMARY:
Erector spinae (ESP) block is a recently described plane block designed to block the dorsal and ventral rami of the thoracic spinal nerves. It is meant to block the ipsilateral trunk. The aim of the study is to demonstrate the efficacy of the ESP block as postoperative analgesia for VATS surgery.

DETAILED DESCRIPTION:
A growing number of thoracic surgeries are performed with a minimally invasive approach called video-assisted thoracoscopic surgery (VATS). VATS has reduced the incision size, the postoperative pain and the morbidity associated with thoracic surgery. Optimal postoperative analgesia for VATS surgery remains an open issue because although it is a lot less painful than a thoracotomy, VATS is a painful procedure with the associated risk of developing chronic pain. Adequate relief leads to early mobilization, potentially improves respiratory functions, and decreases the global stress response secondary to the surgery.

Invasive analgesic techniques such as epidural or paravertebral block for VATS surgery are frequently being replaced for less invasive plane blocks to provide postoperative analgesia. At our center, anesthesiologists tend to perform epidurals only when there is a significant risk of transitioning to an open thoracotomy. Patient controlled analgesia (PCA), remains the usual analgesic technique for VATS surgery at our institution.

Erector spinae (ESP) block is a recently described plane block designed to block the dorsal and ventral rami of the thoracic spinal nerves. It is meant to block the ipsilateral trunk. The aim of the study is to demonstrate the efficacy of the ESP block as postoperative analgesia for VATS surgery.

ELIGIBILITY:
Inclusion Criteria:

• Patients > 18 years old with to ASA status I-III, undergoing VATS for lobectomy or wedge.

Non-inclusion Criteria:

* < 18 years old
* BMI > 35
* Chronic pain history with regular opioid and/or gabapentinoids use during the 2 weeks before surgery
* Regular marijuana use
* History of thoracic surgery on the operated side
* Epidural analgesia preferred due to an anticipated high risk of conversion to thoracotomy
* Unable to communicate with the investigators
* Receiving anticoagulation or experiencing any bleeding disorder
* Surgery for empyema and sympathectomy
* Known allergy to local anesthetics, fentanyl or hydromorphone
* Active infection at injection sites
* Preexisting neurological deficit or psychiatric illness
* Severe cardiovascular disease
* Liver failure
* Renal failure (estimated glomerular filtration rate <15 mL/ min/1.73 m2)
* Pregnancy

Exclusion Criteria:

* Perioperative conversion to thoracotomy
* Severe intra- or postoperative bleeding
* Patients requiring postoperative mechanical ventilation
* Technical inability to proceed with the blocks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Postoperative hydromorphone consumption | 24 hours.
  Using the Patient-Controlled Analgesia pumps, we will be able to calculate the amount of Hydromorphone that will be consumed by patients in each of our intervention arms.

SECONDARY OUTCOMES:
Thorax visual analog pain scores (VAS) : scale 0 (no pain) to 10 (worst) | 1-6-12-18-24 hours.
  Using a regular 1 to 10 visual analog chart, post-surgery.
Total opioid consumption post-surgery | 1-6-12-18-24 hours.
  Using the Patient-Controlled Analgesia pumps, we will be able to calculate the amount of Hydromorphone that will be consumed by patients in each of our intervention arms.
PONV Score : 1 to 3 (1- No nausea, 2- Nausea, 3- Vomiting) | 1-6-12-18-24 hours.
  PONV Score (3 points).
Ramsay Sedation Scale (RSS) 1 to 6 (1- Awake and Agitated, 2- Awake but calm to 6- Asleep and no response to loud auditory stimulus) | 1-6-12-18-24 hours.
  Sedation score of patients : Ramsay Sedation Scale (6 points).
  1. Awake ; agitated or restless or both.
  2. Awake ; cooperative, oriented, and tranquil.
  3. Awake but responds to commands only.
  4. Asleep ; brisk response to light glabellar tap or loud auditory stimulus.
  5. Asleep ; sluggish response to light glabellar tap or loud auditory stimulus.
  6. Asleep ; no response to glabellar tap or loud auditory stimulus.
Global QoR-15 score : 0 to 150 (worst to best) | Pre and postoperatively
  QoR-15 Score is a score concerning the Quality of Recuperation post-surgery containing 15 questions with scales 0 to 10 (worst to best). The same questions are also asked before the surgery to understand the impact of the surgery and anesthesia.
Amount of intraoperative Fentanyl use | Intraoperatively
  Amount in micrograms

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Clairoux, MD, Principal Investigator — Maisonneuve-Rosemont Hospital / CIUSSS de l'Est-de-l'Île-de-Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Protected health information will not be re-used or disclosed to a third party except as required by law, for authorized oversight of the research, or as permitted by an authorization signed by the research subject.

REFERENCES:
- [Background] Alzahrani T. Pain relief following thoracic surgical procedures: A literature review of the uncommon techniques. Saudi J Anaesth. 2017 Jul-Sep;11(3):327-331. doi: 10.4103/sja.SJA_39_17. PMID 28757835
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Forero M, Rajarathinam M, Adhikary S, Chin KJ. Erector spinae plane (ESP) block in the management of post thoracotomy pain syndrome: A case series. Scand J Pain. 2017 Oct;17:325-329. doi: 10.1016/j.sjpain.2017.08.013. Epub 2017 Sep 12. PMID 28919152
- [Background] Hamilton DL, Manickam B. Erector spinae plane block for pain relief in rib fractures. Br J Anaesth. 2017 Mar 1;118(3):474-475. doi: 10.1093/bja/aex013. No abstract available. PMID 28203765
- [Background] Kaplowitz J, Papadakos PJ. Acute pain management for video-assisted thoracoscopic surgery: an update. J Cardiothorac Vasc Anesth. 2012 Apr;26(2):312-21. doi: 10.1053/j.jvca.2011.04.010. Epub 2011 Jun 25. No abstract available. PMID 21705236
- [Background] Kartalov A, Jankulovski N, Kuzmanovska B, Zdravkovska M, Shosholcheva M, Spirovska T, Petrusheva AP, Tolevska M, Srceva M, Durnev V, Jota G, Selmani R, Sivevski A. Effect of Adding Dexamethasone as a Ropivacaine Adjuvant in Ultrasound-Guided Transversus Abdominis Plane Block for Inguinal Hernia Repair. Pril (Makedon Akad Nauk Umet Odd Med Nauki). 2015;36(3):35-41. doi: 10.1515/prilozi-2015-0076. PMID 27442394
- [Background] Khalil AE, Abdallah NM, Bashandy GM, Kaddah TA. Ultrasound-Guided Serratus Anterior Plane Block Versus Thoracic Epidural Analgesia for Thoracotomy Pain. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):152-158. doi: 10.1053/j.jvca.2016.08.023. Epub 2016 Aug 21. PMID 27939192
- [Background] Khoshbin E, Al-Jilaihawi AN, Scott NB, Prakash D, Kirk AJ. An audit of pain control pathways following video-assisted thoracoscopic surgery. Innovations (Phila). 2011 Jul;6(4):248-52. doi: 10.1097/IMI.0b013e31822b2cc1. PMID 22437983
- [Background] Kim DH, Oh YJ, Lee JG, Ha D, Chang YJ, Kwak HJ. Efficacy of Ultrasound-Guided Serratus Plane Block on Postoperative Quality of Recovery and Analgesia After Video-Assisted Thoracic Surgery: A Randomized, Triple-Blind, Placebo-Controlled Study. Anesth Analg. 2018 Apr;126(4):1353-1361. doi: 10.1213/ANE.0000000000002779. PMID 29324496
- [Background] Kosinski S, Fryzlewicz E, Wilkojc M, Cmiel A, Zielinski M. Comparison of continuous epidural block and continuous paravertebral block in postoperative analgaesia after video-assisted thoracoscopic surgery lobectomy: a randomised, non-inferiority trial. Anaesthesiol Intensive Ther. 2016;48(5):280-287. doi: 10.5603/AIT.2016.0059. PMID 28000203
- [Background] Lonnqvist PA, MacKenzie J, Soni AK, Conacher ID. Paravertebral blockade. Failure rate and complications. Anaesthesia. 1995 Sep;50(9):813-5. doi: 10.1111/j.1365-2044.1995.tb06148.x. PMID 7573876
- [Background] Okmen K, Metin Okmen B. Evaluation of the effect of serratus anterior plane block for pain treatment after video-assisted thoracoscopic surgery. Anaesth Crit Care Pain Med. 2018 Aug;37(4):349-353. doi: 10.1016/j.accpm.2017.09.005. Epub 2017 Oct 12. PMID 29033355
- [Background] Scimia P, Basso Ricci E, Droghetti A, Fusco P. The Ultrasound-Guided Continuous Erector Spinae Plane Block for Postoperative Analgesia in Video-Assisted Thoracoscopic Lobectomy. Reg Anesth Pain Med. 2017 Jul/Aug;42(4):537. doi: 10.1097/AAP.0000000000000616. No abstract available. PMID 28632673
- [Background] Steinthorsdottir KJ, Wildgaard L, Hansen HJ, Petersen RH, Wildgaard K. Regional analgesia for video-assisted thoracic surgery: a systematic review. Eur J Cardiothorac Surg. 2014 Jun;45(6):959-66. doi: 10.1093/ejcts/ezt525. Epub 2013 Nov 27. PMID 24288340
- [Background] Taylor R, Massey S, Stuart-Smith K. Postoperative analgesia in video-assisted thoracoscopy: the role of intercostal blockade. J Cardiothorac Vasc Anesth. 2004 Jun;18(3):317-21. doi: 10.1053/j.jvca.2004.03.012. PMID 15232812